CLINICAL TRIAL: NCT05068687
Title: Peroperative Assessment of Tumour Resection Margins Using High-resolution 18F-FDG-PET/CT in Malignancies of the Head and Neck, a Pilot Study
Brief Title: Peroperative Assessment of Malignancies of the Head and Neck Using High-resolution 18F-FDG-PET/CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: XEOS Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BC-05493
Record Dates: First submitted 2021-09-24; First posted 2021-10-06 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2021-09

CONDITIONS: Head and Neck Neoplasms; Thyroid Neoplasm; Skin Neoplasm
MeSH Terms: conditions — Head and Neck Neoplasms; Thyroid Neoplasms; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intraoperative high-resolution PET-CT imaging of resected malignancy (Experimental)
  Interventions: Diagnostic Test: high-resolution PET-CT specimen imaging.

INTERVENTIONS:
Diagnostic Test: high-resolution PET-CT specimen imaging. — Included patients are given a single weight-dependent activity of 18F-FDG at the department of Nuclear Medicine. After administration, patients are brought to the operating room where standard of care surgical removal of the malignancy is performed.
  The resected specimen(s) are brought to the imaging lab and scanned using a preclinical and/or a dedicated specimen PET/CT device. Following PET/CT imaging, the specimen is brought to the department of pathology, where it is sliced. Some of these slices are then rescanned using the preclinical PET/CT device. Moreover, frozen sections are made from one of these slices with macroscopically visible malignant tissue and placed on an autoradiograph overnight. Finally, the imaging results are then correlated to the results found during histopathological analysis of the specimens.

SUMMARY:
In this study, patients diagnosed with a pathology-proven malignancy of the head and neck will receive a routine clinical activity of 18F-FDG ((18)F-luorodeoxyglucose) before undergoing standard of care surgical resection of the malignancy. Following the resection, the 18F-FDG-infused malignancy will be investigated utilizing a novel high-resolution Positron Emission Tomography (PET) and Computed Tomography (CT) scan. Slicing of the malignancy will be followed by additional PET/CT-scanning and autoradiography of the sliced specimen. The results found during image analysis will be compared to the results of the gold standard of histopathology. As this is no approved way of assessing the tumour's margin, the conclusion of the scan will not be used as a method for changing the patients' treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or multiple pathologically proven malignancies in the head and neck region (targeted lesions), independent of origin and stage.
* Patient is planned for the surgical resection of the targeted lesion.
* Age ≥ 18 years.
* Karnofsky performance scale ≥30
* Patient has given informed consent according to the International Conference on Harmonization (ICH) Good Clinical Practice (GCP) guidelines in accordance with the declaration of Helsinki.

Exclusion Criteria:

* Patient is planned for a treatment regimen which does not include standard surgical resection of the targeted lesion.
* Pregnant or actively lactating women.
* Blood glucose level ≥ 200mg/dl or more on the day of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Determine margin status in malignancies of the head and neck | 1 week after administration
  To investigate the ability of high-resolution 18F-FDG-PET/CT-scan to determine the margin status in malignancies of the head and neck. This will be compared to the gold standard of histopathological examination.

SECONDARY OUTCOMES:
Characterize the ideal activity of 18F-FDG | During data-analysis
  The characterization of the ideal dose of 18F-FDG necessary for specimen imaging with a sufficient signal-to-noise ratio. This dose will be identified using post-processing image reconstruction on the specimen resulting from patients given a standard diagnostic activity of 18F-FDG.
Identify positive lymph nodes using 18F-FDG PET/CT | 1 week after administration
  To investigate the ability of high-resolution 18F-FDG-PET/CT to identify positive lymph nodes excised by neck dissection. This will be quantified as sensitivity and specificity compared to the gold standard of histopathological examination.
Correlate distribution of 18F-FDG with histopathology | 1 day after administration
  To correlate the distribution of 18F-FDG in and around tumoral tissue with the histopathology of the specimen. This will be performed by correlating the results obtained from the PET/CT-scan of (sliced) tumoral specimens and autoradiography of a frozen section of the tumour.

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Huvenne, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Result] Debacker JM, Schelfhout V, Brochez L, Creytens D, D'Asseler Y, Deron P, Keereman V, Van de Vijver K, Vanhove C, Huvenne W. High-Resolution 18F-FDG PET/CT for Assessing Three-Dimensional Intraoperative Margins Status in Malignancies of the Head and Neck, a Proof-of-Concept. J Clin Med. 2021 Aug 22;10(16):3737. doi: 10.3390/jcm10163737. PMID 34442033
- [Derived] Debacker JM, Maris L, Cordier F, Creytens D, Deron P, Descamps B, D'Asseler Y, De Man K, Keereman V, Libbrecht S, Schelfhout V, Van de Vijver K, Vanhove C, Huvenne W. Direct co-registration of [18F]FDG uptake and histopathology in surgically excised malignancies of the head and neck: a feasibility study. Eur J Nucl Med Mol Imaging. 2023 Jun;50(7):2127-2139. doi: 10.1007/s00259-023-06153-z. Epub 2023 Mar 1. PMID 36854863